CLINICAL TRIAL: NCT00385645
Title: Comparison of 2 Alternative Antiretroviral Combinations in HIV Post-exposure Prophylaxis: AZT-3TC (Combivir®) + Lopinavir-ritonavir (Kaletra®) Versus AZT-3TC (Combivir®)+ Atazanavir (Reyataz®). Multicentre, Prospective, Randomized, Open Study
Brief Title: Atazanavir or Lopinavir in HIV Post-exposure Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Felipe Garcia Alcaide, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DATEM-PEP
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Combivir+Kaletra
Drug: Combivir+Reyataz

SUMMARY:
The study compares the adherence of 240 HIV-negative subjects randomly assigned to 2 different antiretroviral therapies for 28 days after accidental exposure to HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* HIV exposure requiring prophylaxis under current guidelines

Exclusion Criteria:

* Pregnancy
* Suspected drug resistance in source case
* Contraindications to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2006-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proportions of patients completing 28-day antiretroviral treatment (ARVT)

SECONDARY OUTCOMES:
Proportion of HIV-seropositive at 6 months
Incidence of adverse effects (clinical and laboratory) during ARVT
Adherence to ARVT, time to adherence loss.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Garcia, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (7):
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Joan XXIII, Tarragona, Tarragona

REFERENCES:
- [Derived] Diaz-Brito V, Leon A, Knobel H, Peraire J, Domingo P, Clotet B, Dalmau D, Cruceta A, Arnaiz JA, Gatell JM, Garcia F; DATEMPEP study group. Post-exposure prophylaxis for HIV infection: a clinical trial comparing lopinavir/ritonavir versus atazanavir each with zidovudine/lamivudine. Antivir Ther. 2012;17(2):337-46. doi: 10.3851/IMP1955. Epub 2011 Nov 25. PMID 22293542